CLINICAL TRIAL: NCT06198010
Title: Advancing Safe, Comprehensive, Digitally-Enabled Cancer Pain Management (ASCENT) Clinical Trial - Main
Brief Title: A Collaborative Intervention for Improving Cancer Pain Management in Cancer Survivors (ASCENT)
Acronym: ASCENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ASCENT_MAIN; R33CA278594 (NIH); 23-010838 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm; Hematopoietic and Lymphatic System Neoplasm
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patient Reported Outcome Measures will be administered at baseline by a study coordinator and at 3 and 6 months by a blinded, bilingual, assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (enhanced usual care) (Active Comparator): Patients receive enhanced usual care, which includes access to the educational and pain self-management materials developed for the ASCENT trial (the ASCENT guide).
  Interventions: Other: Best Practice; Other: Educational Intervention; Other: Questionnaire Administration; Other: Electronic Health Record Review
- Arm II (ASCENT intervention) (Experimental): Patients receive the ASCENT guide and attend 3 video or phone calls over 30 minutes each with their CHW and/or PCM. During the first call, patients discuss barriers to receiving help for their pain with their CHW. During the second call, patients work with their PCM to develop an action plan for addressing their pain using the different techniques and interventions detailed in the ASCENT guide. During the third and final call, patients meet with both their CHW and PCM to discuss specialist recommendations for their pain management plan. After the final visit, patients will be contacted by the CHW or PCM every other week to monitor their progress and may also be contacted as-needed based on the their reported pain intensity, symptoms, or reported barriers.
  Interventions: Other: Best Practice; Other: Educational Intervention; Other: Questionnaire Administration; Other: Electronic Health Record Review; Procedure: Health Telemonitoring; Behavioral: Cancer Pain Management

INTERVENTIONS:
Other: Best Practice — Receive enhanced usual care
  Other Names: standard of care; standard therapy
Other: Educational Intervention — Receive ASCENT guide
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Questionnaire Administration — Ancillary studies
Other: Electronic Health Record Review — Ancillary studies
Procedure: Health Telemonitoring — Attend video or phone calls with a CHW and/or PCM
  Arms: Arm II (ASCENT intervention)
Behavioral: Cancer Pain Management — Receive personalized pain management plan
  Other Names: management of cancer pain
  Arms: Arm II (ASCENT intervention)

SUMMARY:
This clinical trial tests a collaborative pain management intervention (ASCENT) for improving cancer pain in cancer survivors. Cancer pain is prevalent, under-treated, and remains a major cause of suffering, impairment, and disability for millions of Americans. Individual pain interventions and care models show promise for cancer pain in controlled settings. All cancer survivors stand to benefit from electronic health record innovations, as they can experience profound pain outcomes, including marked under- and over-prescribing of opioids. Digitally facilitated solutions are especially helpful and can be customized to address patient needs. The ASCENT intervention provides patients with an educational guide that describes techniques for addressing cancer pain, and uses community health workers and pain care managers to coach patients through a personalized pain management plan. This study may help researchers learn how pain management strategies can improve cancer pain and lower risk of opioid exposure and dependency in cancer survivors.

DETAILED DESCRIPTION:
NOTE: Although Mayo Clinic in Arizona, Mayo Clinic in Florida, and Mayo Clinic in Rochester are the main study locations, this study is also recruiting (enrolling remotely) at the following Mayo Clinic Health System locations. The study is virtual/remote, so no travel is required.

Mayo Clinic Health Systems-Mankato Mankato, MN 56001, US

Mayo Clinic Health System in Albert Lea Albert Lea, MN 56007, US

Mayo Clinic Health System in Austin Austin, MN 55912, US

Mayo Clinic Health System-Eau Claire Clinic Eau Claire, WI 54701, US

Mayo Clinic Health System-Franciscan Healthcare La Crosse, WI 54601, US

PRIMARY OBJECTIVE:

I. To test a validated collaborative care model-based intervention aimed at improving pain control among cancer survivors by promoting multimodal pain care (MMPC) to reduce inappropriate opioid use and by addressing social determinants of health (SDOH) that impede a patient's access to appropriate care.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive enhanced usual care, which includes access to the educational and pain self-management materials developed for the ASCENT trial (the ASCENT guide).

ARM II: Patients receive the ASCENT guide and attend 3 video or phone calls over 30 minutes each with their community health worker (CHW) and/or pain care manager (PCM). During the first call, patients discuss barriers to receiving help for their pain with their CHW. During the second call, patients work with their PCM to develop an action plan for addressing their pain using the different techniques and interventions detailed in the ASCENT guide. During the third and final call, patients meet with both their CHW and PCM to discuss specialist recommendations for their pain management plan. After the final visit, patients will be contacted by the CHW or PCM every other week to monitor their progress and may also be contacted as-needed based on the their reported pain intensity, symptoms, or reported barriers.

ELIGIBILITY:
Inclusion Criteria:

* A qualifying liquid or solid cancer diagnosis with visits at a participating Mayo site in the past 15 years

  * Including malignant hematology

    * Lymphoma
    * Myeloma
    * Chronic leukemias
* Age >= 18
* Numeric Rating Scale (NRS) pain score of >= 5/10
* Pain that developed or worsened following cancer diagnosis
* Fit the description of either rural or Hispanic or both

Exclusion Criteria:

* Patient Health Questionnaire - 8 (PHQ8) score of >= 13
* Hospice enrollment
* Skilled nursing facility, inpatient rehabilitation facility, or long-term care placement
* Encounters with Palliative Care or the Pain Clinic in the past two months or upcoming two months
* Any mention of hospice referral in medical oncology encounter notes (assess through textual search of the Mayo Data Explorer)
* Affirmative response to, "Are you usually confined to a bed or chair more than a third of your waking hours because of your health?"
* Currently homeless
* Do not feel safe in their home
* New or worsening chest pain, chest tightness, or chest pressure
* Back pain that is associated with a new or worsening weakness, control of bowels/bladder, or difficulty walking
* Lightheadedness, inability to keep down food or fluids, or vomiting blood or dark coffee-grounds-like material
* New or worsening headaches that are associated with vision changes, nausea, balance issues, or problems with speech
* Screens positive for use of non-cannabis drug use a a frequency of monthly or greater
* Inability to engage with the intervention due to medical or psychological response

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Score | Baseline, 3 months, 6 months
  Will be measured using the Brief Pain Inventory Short Form (BPI SF), a 4-item questionnaire answered on a scale from 0 (no pain) to 10 (pain as bad as you can imagine). A higher score indicates worse pain.

SECONDARY OUTCOMES:
Physical function | Baseline, 3 months, 6 months
  Will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Functioning Short Form (SF) 6b, a 6-item questionnaire that measures the effects of pain on physical functioning over the past 7 days. Questions are answered on a scale of 1-5, with higher scores indicating more pain interference.
Perceived Quality of Life | Baseline, 3 months, 6 months
  Will be measured using the European Quality of Life 5 Dimensions 3 Level (EQ-5D-3L) questionnaire, which measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each component has three response levels of severity: no problems, some problems, extreme problems.
Depression | Baseline, 3 months, 6 months
  Will be measured using the Patient Health Questionnaire-2 (PHQ-2), a two-item questionnaire answered with responses from 0 (not al all) to 3 (nearly every day). A higher score indicates a higher level of depression.
Anxiety | Baseline, 3 months, 6 months
  Will be measured using the Generalized Anxiety Disorder-2 (GAD-2) scale, a two-item questionnaire answered with a score of 0 (not at all) to 3 (nearly every day). A higher score indicates higher frequency of being bothered by anxiety.
Sleep | Baseline, 3 months, 6 months
  Will be measured using the PROMIS Sleep Disturbance 6a, a 6-item questionnaire assessing sleep disturbance over the past 7 days. Each question is answered with a score of 1-5, with a higher score indicating greater sleep disturbance.
Employment status | Baseline, 3 months, 6 months
  Employment status will be self-reported
Adherence to behavioral multimodal pain care plan components | Baseline, 3 months, 6 months
  Will be measured using logged count data.
Use of study electronic-tools | Baseline, 3 months, 6 months
  Will be measured in minutes/week that participants access available electronic tools.
Social isolation | Baseline, 3 months, 6 months
  Will be measured using the PROMIS SF 4a, a six-item questionnaire with each question answered on a five-point scale from 1 (never) to 5 (very often). Higher scores indicate greater perceived social isolation.
Opioid consumption | Up to 6 months
  Will be measured in oral morphine equivalents and collected using electronic health record (EHR) prescriptions.
Health care utilization | Up to 6 months
  Will be measured by reviewing the electronic health record (EHR) and administrative billing data for incidents of hospitalization and emergency department visits

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L. Cheville, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials